CLINICAL TRIAL: NCT03602235
Title: High Dose Ascorbic Acid (HDAA) in Patients With Plasma Cell Disorders
Brief Title: High Dose Ascorbic Acid for Plasma Cell Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christopher Strouse (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Christopher Strouse, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201804754
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Ascorbic Acid; Injections; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Low dose melphalan + high dose ascorbate acid (HDAA) (Experimental): Patients will receive a test dose of 15g of HDAA prior to starting treatment dose. This will be mainly to rule out allergic reactions.
  HDAA + Melphalan:
  HDAA on day 1 and day 4 in combination with melphalan 12.5 mg/m2, followed by 2 additional doses of HDAA on day 2 and day 5.
  A 3 + 3 cohort method will be used for this study. After successfully completing the test dose, subjects will receive 50gms, 75gms and 100gms of ascorbate per infusion in 3 different cohorts. Dose modifications are not made for weight or body surface area.
  Interventions: Other: Ascorbate; Drug: Melphalan

INTERVENTIONS:
Other: Ascorbate — Ascorbate is in the vitamin drug class
  Other Names: Ascorbate Acid; Ascorbic Acid for Injection, USP
Drug: Melphalan — Melphalan is an alkylating agent coupled to an amino acid
  Other Names: L-phenylamine mustard; L-PAM; L-Sarcolysin

SUMMARY:
This is a Phase I single-arm open-label clinical study primarily assessing the safety and secondarily, the relative efficacy of low dose melphalan + high dose ascorbate acid (HDAA) in relapsed refractory patients with multiple myeloma.

DETAILED DESCRIPTION:
This is a phase 1 study for patients with relapsed refractory multiple myeloma. Patients will receive a 15-gram test dose, and a maximum of 3 cycles, each composed of 4 doses of high-dose ascorbic acid (HDAA) and 2 doses of melphalan. This study will enroll 9 patients with relapsed refractory multiple myeloma. The starting dose of ascorbic acid will be 50 grams. Using a 3+3 dose escalation, the dose will potentially increase to 75 grams then 100 grams.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Diagnosis of multiple myeloma per IMWG criteria(26)
* Patients must have progressive disease following 3 or more prior lines of therapy.

  * Prior treatment must include a proteasome inhibitor, an immunomodulatory agent (IMiD), and an anti-CD38 monoclonal antibody.
  * Patients must not be candidates for regimens known to provide clinical benefit in relapsed or refractory multiple myeloma based on the investigator's judgement.
  * If a patient declines such therapy, this must be recorded in the study files. 4. Subjects must have measurable disease, including at least one of the criteria below:
  * SPEP demonstrating M-protein quantities ≥ 0.5 g/dl
  * UPEP demonstrating monoclonal protein ≥ 200 mg/24hr
  * Involved serum free light chain levels > 100 mg/L and an abnormal kappa/lambda (κ/λ)ratio
  * For patients with immunoglobulin class A (IgA) myeloma whose disease can only be reliably measured by quantitative immunoglobulin measurement, a serum IgA level ≥ 500 mg/dl will qualify as measurable disease
  * Non-secretory participants are eligible provided the participant has > 20% bone marrow plasmacytosis
* Adequate organ function:

  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L without growth factor support for 7 days
  * Platelets (plt) ≥ 50 x 10^9/L without transfusion for 7 days.
  * Hemoglobin ≥ 8.0 g/dl, transfusion support permitted
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3.0x upper limit of normal (ULN)
  * Serum bilirubin ≤ 1.5 x ULN
  * Estimated serum creatinine clearance of ≥ 45 mL/min using the Cockcroft-Gault equation or directly calculated from the 24-hour urine collection method.
  * International normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) < 1.5 x ULN
  * Left Ventricular Ejection Fraction by ECHO or MUGA of ≥ 40%.
  * Participants must have a performance status of 0-2 based on ECOG criteria.
  * For people of child bearing potential negative serum or urine pregnancy test (sensitivity of at least 25 mIU/mL) at screening

Exclusion Criteria

* Known hypersensitivity or allergy to ascorbic acid or melphalan
* Participants must not have a concurrent malignancy unless it can be adequately treated by non- chemotherapeutic intervention. Participants may have a history of prior malignancy, provided they have not had any chemotherapy within 365 days of study entry AND their life expectancy exceeds 5 years with respect to the concurrent malignancy at the time of study entry.
* Participants must not have life-threatening comorbidities.
* Known human immunodeficiency virus(HIV) disease (requires negative test for clinically suspected HIV infection).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, recent (within 6 months) myocardial infarction, uncontrolled or symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension on appropriate therapy or psychiatric illness/social situations that would limit compliance with study requirements.
* Concurrent use of Coumadin (warfarin)
* Patients with G6PD deficiency
* Patients with a history of oxalate renal stones or a known history of multiple renal stones
* Diabetic patients who rely on a glucometer to dose insulin as ascorbate can interfere with glucometer readings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Number of treatment related adverse events as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 | First day of treatment through 28 days
  Adverse events occuring within the DLT assessment window which do not resolve in less than 72 hours and are not clearly and incontrovertibly due to extraneous causes.

SECONDARY OUTCOMES:
Rate of minimal residual disease (MRD) negativity through bone marrow testing and imaging | Through 28 days after the end of treatment
  MRD will be determined by highly sensitive, eight color flow on bone marrow sample. Functional imaging, such as PET scan and MRI will also be performed to assess the disease status.
Overall response rate based on International Myeloma Working Group (IMWG) criteria | Through 24 months after the end of treatment
  Response to treatment will be assessed by IMWG criteria.
Categorize and quantify adverse events compared to historical control | Up to 24 months following the end of treatment for the last patient
  The number and severity of all adverse events will be summarized by simple descriptive statistics and compared to a historical control.
Oxidative stress parameters in plasma through blood testing | Through 24 months after the end of treatment
  Blood will be drawn and serum iron, TIBC, serum ferritin and transferrin saturation levels tested.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Strouse, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No